CLINICAL TRIAL: NCT02126891
Title: FACEFI : Cardiac Fatigue During Intense Exercises - Pilot Study
Acronym: FACEFI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 2013-A01524-41
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-04

CONDITIONS: Muscle; Fatigue, Heart
Keywords: Cardiac functions; Endurance training; Senior athletes
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Canoeists (Experimental): 13 canoeists from a training center of the French canoeing team
  Interventions: Procedure: Tests
- Military (Experimental): 10 young recruits in military school of officers in ground forces of the French army
  Interventions: Procedure: Tests

INTERVENTIONS:
Procedure: Tests — Individual parameters of echocardiography and heart rate variability

SUMMARY:
To attest if a cardiac fatigue appears (and to measure it if it does) during intense physical exercises in two groups of subjects:

* Canoeists from a training center of the French canoeing team during an intensive session of three weeks of endurance training;
* Young recruits in military school of officers in ground forces of the French army during an intensive.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men between 18 and 35 years old;
* Giving their writing informed consent;
* And affiliated to the French social security.

Exclusion Criteria:

* To be a smoker.
* To present any known pathology that forbids the realisation of any test, or that can alter the measurements: cardiovascular risk factors treated or not (diabetes, dyslipidaemia, arterial hypertension, obesity), cardiac arrhythmia, coronary disease, heart failure, cardiac pacemaker or defibrillator, valvular disease after surgery or not, kidneys failure with dialyse or not, kidney pulmonary cardiac or liver transplantation, chronic bronchopneumopathy, asthma, etc.
* To take any medication that could alter autonomic nervous system or cardiovascular adaptation to maximal exercise (anti-arrhythmia, anti-hypertensive, anti-inflammatory,…).
* Drinking exciting drinks (coffee or tee for example) in the 12h before the tests.
* To be under legal protection (trusteeship, guardianship) or to be deprived of liberty.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Measure of classical echocardiographic parameters to attest systolic and diastolic functions | day 8 (canoeists) / day 5 (military)
  Speckle tracking will also be used to get strain parameters of the left ventricle. Measure will by recording daily before, during, and after a period of intensive training, in order to attest possible cardiovascular effects of such periods.
  Echocardiographic data will be recorded at rest and during a submaximal exercise.

SECONDARY OUTCOMES:
Measure of classical heart rate variability parameters | day 8 (canoeists) / day 5 (military)
  Measure will by recording daily before, during, and after a period of intensive training, in order to attest possible cardiovascular effects of such periods.
  Measure will be recorded during 5 min resting and 5 min standing.

CONTACTS AND LOCATIONS:
Overall Officials: François FC Carré, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France